CLINICAL TRIAL: NCT03083106
Title: Snoring Intervention Via Elevoplasty in a Non-surgical Clinical Environment
Acronym: SILENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zelegent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCP002-001
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2017-03

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Intervention Model Description: Single Group Compared to Baseline, Non-Randomized, Multi-Center, Prospective Safety & Efficacy Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Elevoplasty treatment (Other): Single Group Compared to Baseline, Non-Randomized, Multi-Center, Prospective
  Interventions: Device: Elevoplasty

INTERVENTIONS:
Device: Elevoplasty — The Elevo™ Kit Snoring Intervention Device is designed to facilitate deployment of the Elevo™ suture implant into the submucosal tissue of the soft palate via a minimally invasive, outpatient procedure performed by an otolaryngologist in a medical office setting.

SUMMARY:
Single Group Compared to Baseline, Non-Randomized, Multi-Center, Prospective Safety & Efficacy Study

DETAILED DESCRIPTION:
Evaluate the safety and efficacy of the Zelegent, Inc. Elevo™ Kit Snoring Intervention Device (a minimally invasive, barbed, absorbable suture implant) in the reduction of simple snoring through subjective evaluation of snoring and objective snoring sound analysis.

The Zelegent, Inc. Elevo™ Kit Snoring Intervention Device is intended to reduce or eliminate simple snoring in the target patient population via minimally invasive implantation of specialized barbed, absorbable sutures in the soft palate for the purpose of stiffening by way of shortening and lifting the soft palate thereby addressing the root cause of snoring.

ELIGIBILITY:
Inclusion Criteria:

* Age > 22 years (no maximum age)
* Has consistent Bed/Sleep Partner willing to provide Co-Participant Informed Consent
* Apnea Hypopnea Index (AHI) of < 15 verified by polysomnogram (PSG) or by SNAP® Diagnostics Home Sleep Study (HSS)
* Has basic computer literacy (e.g., email) and home internet access or smartphone
* Chronic, simple snoring (verified by Bed/Sleep Partner)
* No prior surgical treatment for snoring
* Bed/Sleep Partner willing and capable of providing Informed Consent

Exclusion Criteria:

* Age < 22 years
* Has no consistent Bed/Sleep Partner
* Apnea Hypopnea Index (AHI) > 15 indicative of Obstructive Sleep Apnea
* Intermittent or occasional snoring
* Body Mass Index (BMI) > 32 kg/m2
* Modified Mallampati 3 or 4
* Tonsil Grade 3 or 4+
* Significant nasal obstruction
* Previous palatal surgery
* Current cigarette smoker
* Known history of coronary artery disease or stroke
* Chronic obstructive pulmonary disease (COPD)
* Diabetes (Type I or Type II) non-controlled by medical management
* Major depression or non-controlled psychiatric illness
* Drug or alcohol abuse
* Untreated or poorly controlled hypertension
* Anticoagulation therapy
* History of bleeding or clotting disorder
* Pregnant Female

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Mean within-subject change in Snoring Visual Analog Scale from pre-treatment with the device ("Elevo Kit") to Snoring Visual Analog Scale post-treatment with the device ("Elevo Kit"). | Thirty (30) days post device intervention
  Difference between the two following parameters: (1) Snoring Visual Analog Scale (VAS) pre-intervention with the device ("Elevo Kit") (2) Snoring Visual Analog Scale (VAS) post-intervention with the device ("Elevo Kit"). Resulting value is in an absolute number i.e., a numeric 1 to 10 response by the sleep/bed partner to the VAS inquiry "Please indicate, by selecting a number on the scale below, the loudness of your partner's snoring." A numeric "0" response corresponds to "Light Loudness". A numeric "5" response corresponds to "Moderate Loudness". A numeric "10" response corresponds to "Intense Loudness".

SECONDARY OUTCOMES:
Mean within-subject change in Snoring Visual Analog Scale from pre-treatment with the device ("Elevo Kit") to Snoring Visual Analog Scale post-treatment with the device ("Elevo Kit"). | Ninety (90) days post device intervention
  Difference between the two following parameters: (1) Snoring Visual Analog Scale (VAS) pre-intervention with the device ("Elevo Kit") (2) Snoring Visual Analog Scale (VAS) post-intervention with the device ("Elevo Kit"). Resulting value is in an absolute number i.e., a numeric 1 to 10 response by the sleep/bed partner to the VAS inquiry "Please indicate, by selecting a number on the scale below, the loudness of your partner's snoring." A numeric "0" response corresponds to "Light Loudness". A numeric "5" response corresponds to "Moderate Loudness". A numeric "10" response corresponds to "Intense Loudness".
Mean within-subject change in Snoring Visual Analog Scale from pre-treatment with the device ("Elevo Kit") to Snoring Visual Analog Scale post-treatment with the device ("Elevo Kit"). | One hundred eighty (180) days post device intervention
  Difference between the two following parameters: (1) Snoring Visual Analog Scale (VAS) pre-intervention with the device ("Elevo Kit") (2) Snoring Visual Analog Scale (VAS) post-intervention with the device ("Elevo Kit"). Resulting value is in an absolute number i.e., a numeric 1 to 10 response by the sleep/bed partner to the VAS inquiry "Please indicate, by selecting a number on the scale below, the loudness of your partner's snoring." A numeric "0" response corresponds to "Light Loudness". A numeric "5" response corresponds to "Moderate Loudness". A numeric "10" response corresponds to "Intense Loudness".

OTHER OUTCOMES:
Mean within-subject change in SNAP Diagnostics Home Sleep Study (HSS) Measure #1 from pre-treatment with the device ("Elevo Kit") to post-treatment with the device ("Elevo Kit"). | Thirty (30) days post device intervention
  Difference between the two following parameters: (1) Percent (%) of snoring events comprised of the sum of types (I + II) and comprised of the sum of types (III + IV + WL) pre-treatment (2) Percent (%) of snoring events comprised of the sum of types (I + II) and comprised of the sum of types (III + IV + WL) post-treatment.
  Key to Snoring Event Types (as categorized by SNAP Diagnostics, Inc.) Type I: Mostly Palate Type II: Mostly Palate + tongue Type III: Sound, but no particular pattern, can originate from lungs or from upper airway Type IV: High pitch, more diffuse, similar to asthma Type WL: Wheezing-like. Resulting value of Measure #1 is in percents (%). Note: Measure #1 will be repeated via Home Sleep Study at Day 90 post-treatment and will be repeated via Home Sleep Study at Day 180 post-treatment.
Mean within-subject change in SNAP Diagnostics Home Sleep Study (HSS) Measure #2 from pre-treatment with the device ("Elevo Kit") to post-treatment with the device ("Elevo Kit"). | Thirty (30) days post device intervention
  Difference between the two following parameters: (1) Average loudness ratio (loudness is measured in decibels [dB]) of events comprised of the sum of types (I + II) and comprised of the sum of types (III + IV + WL) pre-treatment (2) Average loudness ratio of events comprised of the sum of types (I + II) and comprised of the sum of types (III + IV + WL) post-treatment.
  Key to Snoring Event Types (as categorized by SNAP Diagnostics, Inc.) Type I: Mostly Palate Type II: Mostly Palate + tongue Type III: Sound, but no particular pattern, can originate from lungs or from upper airway Type IV: High pitch, more diffuse, similar to asthma Type WL: Wheezing-like. Resulting value of Measure #2 is an absolute number. Note: Measure #2 will be repeated via Home Sleep Study at Day 90 post-treatment and will be repeated via Home Sleep Study at Day 180 post-treatment.
Mean within-subject change of Pittsburgh Sleep Quality Index (PSQI) from pre-treatment with the device ("Elevo Kit") to post-treatment with the device ("Elevo Kit"). | Thirty (30) days post device intervention
  Difference between the two following parameters: (1) PSQI Score pre-treatment (2) PSQI Score post-treatment. Resulting value is an absolute number. The PSQI is a self-report (i.e., patient-reported outcome) questionnaire that is comprised of nineteen (19) individual items that create seven (7) components that produce one (1) global score. The PSQI takes 5 - 10 minutes to complete. Note: the PSQI questionnaire will be repeat-administered at Day 90 post device intervention and will be repeat-administered at Day 180 post device intervention.
Mean within-subject change of Epworth Sleepiness Scale (ESS) from pre-treatment with the device ("Elevo Kit") to post-treatment with the device ("Elevo Kit"). | Thirty (30) days post device intervention
  Difference between the two following parameters: (1) ESS Score pre-treatment (2) ESS Score post-treatment. Resulting value is an absolute number. The ESS is a self-report (i.e., patient-reported outcome) scale that is intended to measure daytime sleepiness and that is measured by use of a very short questionnaire. Note: the ESS questionnaire will be repeat-administered at Day 90 post device intervention and will be repeat-administered at Day 180 post device intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Catalano, MD, Principal Investigator — St. Elizabeth's Medical Center
Locations (6):
- United States (6):
  - Entrust Medical Group, Orange, California
  - ChicagoENT (*Note: it's important to capitalize the "ENT"), Chicago, Illinois
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Park Avenue Sinus & Sleep Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will remain confidential to the Investigators and to the Sponsor